CLINICAL TRIAL: NCT07359222
Title: A Clinical Investigation to Validate the Safety and Efficacy of a Nutritional Medical Food Utilized Prior to Surgery to Reduce Post-surgical Complications.
Brief Title: Vis Pre Surgery Medical Food Validation Study
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Frustrations around administrative issues at the study site.
Sponsor: TM Nutrition LLC (Industry)
Collaborators: National University of Natural Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: JSSMC/IEC/18122023/20
Record Dates: First submitted 2025-12-10; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pre-surgical Anxiety; Blood Glucose Concentration; Blood Cortisol Levels; Electrolyte Levels; HbA1c; Surgical Infections; Wound Healing Time; Hospital Stay Time; Readmittance Rate; Mortality
Keywords: Medical food; Pre-surgical medical food

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-treatment control (No Intervention): Usual care
- Vis Pre-Surgery (Experimental): Received Vis Pre-Surgery drink
  Interventions: Other: Pre-surgical medical food

INTERVENTIONS:
Other: Pre-surgical medical food — Vis Pre-Surgery Medical Food
  Arms: Vis Pre-Surgery

SUMMARY:
A pre-market, confirmatory, prospective, interventional, clinical investigation to confirm the clinical safety and performance profile of Vis Pre-surgeryTM that the medical food will reduce pre and post-surgical complications including pre-operative anxiety, infections, hyperglycemia, adrenal insufficiency, post operative nausea and vomiting, decrease wound healing time, decrease length of hospital stay and readmittance and surgical mortality.

DETAILED DESCRIPTION:
In the US alone, 48 million surgeries are performed: 310 million worldwide. Surgical site infections are the most prevalent and deadly post-surgery infection leading to an average of 6% of readmissions costing $10 billion dollars and 400,000 extra hospital days each year. If a surgical site infection occurs, the patient is 42% more likely to die following surgery. If that patient is a diabetic their chance of death increases by five times. Current protocol accepts surgical complications such as infections as known issues that are treated with antibiotic prior to surgery. Surgeons and hospital administrators need a way to affect a positive change in outcomes that augments current procedure and enhances positive outcomes including lowering surgical costs, reducing readmissions, improving hospital scorecards, and increasing survival.

VIS Pre-surgery addresses the specific metabolic and biochemical needs of an adult surgery patient in stress response. Support of these processes with carefully calibrated nutrient therapy reduces the risk of a patient succumbing to infections, especially surgical site infections, urinary tract infections and pneumonia. Product mechanism of action promotes balance of blood sugar levels, an important driver in the infection process while supporting critical immune system requirements to prevent tissue degradation.

This is a pre-market, safety, efficacy, validation clinical investigation to confirm the clinical safety and performance profile of VIS Pre-surgeryTM i. e that the medical food decreases pre-and post-surgical complications while reducing length of hospital stay, readmittance and mortality from surgery with no side effects.

The product is a FDA Medical Food formulated from GRAS (Generally Regarded As Safe) ingredients. The second aspect of the intended purpose (claim) of the medical food is currently supported by the specifications of the individual ingredients. This as clinical claim that can give clinical benefit by applying the cellular method of action for each nutrient, trace mineral and complex carbohydrate.

Patients who are scheduled for elective invasive surgery of upper, lower or cardiothoracic surgery will be asked to participate in the investigation by ingesting VIS Pre-surgery powder dissolved in water the evening prior to surgery at bedtime and again at 4 hours prior to scheduled surgery. Patients will be asked to complete questionnaires, provide blood samples prior to, during and post operatively, submit to abdominal ultrasound, observation and answer questions from coordinators.

Additional data points will be extrapolated from the collection of routine data such as hospital stay time, readmittance and mortality.

Patients will be identified by the PI and Co PIs.

ELIGIBILITY:
Inclusion Criteria:

* adults (≥18 years) scheduled for elective abdominal, cardiac/thoracic, gynecological, or orthopedic surgery

Exclusion Criteria:

* kidney or liver disease, participation in a different clinical investigation that may affect the safety or performance of the investigation, being employees or family members of anyone involved in the investigation, and any other condition or treatment making a subject unsuitable for participation as judged by the Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Adverse events attributable to the study product | Enrollment to 90 day follow up

SECONDARY OUTCOMES:
Postoperative nausea and vomiting (PONV) incidence | From enrollment to 48 hours post-op
30-day hospital readmission | From enrollment to 30 days post-op
Post-operative infections | From enrollment to 90 day follow up

OTHER OUTCOMES:
Blood glucose concentration | Pre-op, peri-op, 24 hours post op, 48 hours post op
HbA1c | Pre-op and 90 days post-op.
Electrolytes | 1 Day Post-op
  sodium, potassium, chloride, calcium, magnesium
Stress hormone | 1 Day Pre-op and 1 Day post-op
  Cortisol
Post-op pain | 1 Day Post-op
  Scale from 0-10
Pre-op emotional state | 1 Day Pre-op
  A single-choice between calm, relaxed, content, tense, worried, upset

CONTACTS AND LOCATIONS:
Overall Officials: Thea Marx, ND, Principal Investigator — TM Nutrition
Locations (1):
- JSS Medical College, Mysuru, India

IPD SHARING:
Plan to Share IPD: No